CLINICAL TRIAL: NCT04332354
Title: Evaluation by CGMS (Continuous Glucose Monitoring System) of the Evolution of the Glycemic Profile in Diabetic Patients in Immediate Post-operative Bariatric Surgery: An Observational Study in Routine Care
Brief Title: Glycemic Profile by CGMS in Diabetic Patients After Bariatric Surgery
Acronym: CGM-BARIA
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: CHU 20-501
Record Dates: First submitted 2020-03-31; First posted 2020-04-02 (Actual); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: Type 2 Diabetes Mellitus in Obese; Bariatric Surgery Candidate
Keywords: continuous glucose monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- T2D diabetes obese subjects: Patients have T2D diabetes and are candidates for bariatric surgery. They will receive routine cares and follow-up and will have CGM measurement before and 2 weeks following the surgery
  Interventions: Other: routine care. No intervention

INTERVENTIONS:
Other: routine care. No intervention — no intervention

SUMMARY:
The aim of this observational prospective monocentric study is to examine glycemic patterns in adult T2D patients candidates to bariatric surgery, by using a continuous glucose monitoring (CGM) sensor over 14 days post-surgery, in order to search for indicators predicting T2D remission 1 year after surgery.

DETAILED DESCRIPTION:
In this exploratory monocentric study performed at the Caen University Hospital in France, adult T2D patients consecutively enrolled for metabolic surgery will be prospectively included for continuous glucose monitoring (CGM) recordings during the month preceding bariatric surgery and during the 2 weeks following surgery. Changes in body weight will be evaluated using weight measurement, BMI measurement and the percentage of excess weight loss (% EWL), calculated using the formula: initial weight-actual weight/initial weight - (25 x height2). Changes in diabetic status will be evaluated by HbA1c assay and collection of data on anti-diabetic treatment maintained during the follow-up. The Ad-Diarem score for predicting diabetes remission will be calculated in each patient from several variables including age, diabetes duration, insulin use, other glucose-lowering agents used, number of glucose-lowering agents used and HbA1c level. The variables recorded by CGM will include : mean daily interstitial glucose concentration (mg/dL), standard deviation (SD) of glucose concentration (mg/dL), coefficient of variation (CV) of glucose concentration corresponding to the SD-to-mean daily interstitial glucose ratio, time in normoglycemia (ie in the stringent 70-140mg/dL target which better reflects normoglycemia than the 70-180 mg/dl target) or time in range (TIR) as a percentage over 24h, time spent in hyperglycemia (ie >140mg/dL) or time above range (TAR) as a percentage over 24h, and time spent in hypoglycemia (<70mg/dL) or time below range (TBR) as a percentage over 24h.

Judgement criteria are defined as follows: the success of bariatric surgery will be defined as a % EWL >50%; normalization of glycemia will be defined as a mean 24-hr interstitial glucose level <100mg/d during the CGM recording period; diabetes remission after metabolic surgery will be defined as an HbA1c level at 1 year after surgery of < 6.0% without the use of any glucose-lowering agent. Such thresholds were chosen to meet the definition of complete remission by the American Society for Metabolic and Bariatric Surgery and the American Diabetes Association.

Quantitative variables will be expressed as mean + standard deviation. Qualitative variables will be expressed as percentages. Differences in quantitative variables, when compared to the pre-operative period, will be examined using Students t-test for paired data or with ANOVA. Analysis of subgroups will be carried out using Chi-2 test. Identification of predictive factors for diabetes remission will be based on analysis of ROC curves and the calculation of area under the curve data, sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV), positive and negative likelihood ratio (LR+ and LR-) at different thresholds for each study variable including the pre-operative and post-operative CGM variables and the Add-Diarem score.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes and obesity (BMI> 35)
* treated with oral anti-diabetic medication and/or insulin therapy
* candidate for bariatric surgery

Exclusion Criteria:

* refusal of CGM recordings
* refusal of bariatric surgery

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: T2D, obesity (BMI>35), candidates for metabolic surgery oral or injectable anti diabetic treatments including insulin injections or pump therapy
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2016-03-30 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
glycemic profile after bariatric surgery | 4-14 days recordings
  CGM recordings 4-14 days of the immediate postoperative period

SECONDARY OUTCOMES:
glycemic profile before bariatric surgery | 5 days recordings
  CGM recordings before bariatric surgery
identification of predictive factors for diabetes remission 1 year after surgery | 5 days recordings for CGM
  CGM variables and Add-Diarem score

IPD SHARING:
Plan to Share IPD: No